CLINICAL TRIAL: NCT06645405
Title: Segmentation and Modeling for Accurate Reconstruction of CT Angiography of Intracranial Large Vessel Occlusion with Artificial Intelligence: a Stepped-wedge, Cluster-randomized Controlled Trial
Brief Title: AI-Driven CTA Reconstruction for Intracranial LVO
Acronym: SMART-AI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, MD, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: SMART-AI
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke; Artificial Intelligence (AI); Endovascular Thrombectomy; CT Angiography
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No AI reconstruction
- AI software (Experimental): An AI approach will be used for automated segmentation and reconstruction of CTA for intracranial LVO. Physicians begin to receive reconstructions and have the authority to view AI-activated images. Diagnosis and treatment decisions will be based on the clinical evaluation and review of the images by the treating physician, as per routine standard of care.
  Interventions: Behavioral: AI algorithm

INTERVENTIONS:
Behavioral: AI algorithm — Artificial intelligence algorithms in the automated reconstruction of intracranial large vessel occlusion (LVO)
  Other Names: AI approach
  Arms: AI software

SUMMARY:
Acute ischemic stroke (AIS) caused by intracranial large vessel occlusion (LVO) in the anterior circulation significantly contributes to stroke-related disability and mortality. Recent randomized controlled trials have demonstrated substantial benefits of endovascular thrombectomy (EVT) when patients are appropriately triaged beforehand. However, accurately orienting the 'missed segment' during EVT remains challenging. Guide-wires often fail to navigate through the occlusion or are mistakenly directed into the small tranches or even cause vessel rupture. To address this clinical need, the investigators developed an artificial intelligence (AI) algorithm to automate the reconstruction of CT angiography (CTA), focusing on the occluded LVO segment. To evaluate the clinical utility of this AI algorithm, the investigators propose a prospective, stepped-wedge cluster-randomized study to determine whether integrating our AI algorithm into AIS care flow can reduce the time for first pass of the thrombus by improving the visualization of the occluded segment on CTA. Physicians will assess patient eligibility for thrombectomy, and all selected patients will receive standard care according to current guidelines. This approach is expected to enhance patient treatment outcomes for endovascular thrombectomy by leveraging readily available data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older.
2. Patients who present with signs and/or symptoms concerning acute ischemic stroke.
3. Patients who undergo noncontrast CT and CT angiography imaging.
4. Patients determined to have an intracranial large vessel occlusion (including the internal carotid artery, middle cerebral artery M1 segment, and M2 segment), and eligible for endovascular treatment.

Exclusion Criteria

1) CT imaging with severe motion artifacts.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AFAT | Immediately after EVT
  The time from target angiography to the initiation of first thrombectomy attempt (angiography-to-first-attempt time [AFAT])

SECONDARY OUTCOMES:
PRT | Immediately after EVT
  The time from groin puncture to final arterial recanalization (puncture-to-recanalization time [PRT])
IPT | Immediately after EVT
  The time from the completion of imaging to the initiation of EVT (imaging-to-puncture time [IPT])
IRT | Immediately after EVT
  The time from imaging completion to final arterial recanalization (imaging-to-recanalization time [IRT])
The rate of successful flow restoration immediately after EVT | Immediately after EVT
  The rate of successful flow restoration immediately after EVT
The rate of symptomatic intracerebral hemorrhage within 24 hours post-EVT | 24 hours post-EVT
  The rate of symptomatic intracerebral hemorrhage within 24 hours post-EVT
The rate of procedure-related complications | Immediately after EVT
  The rate of procedure-related complications
The rate of functional independence at 90 days post-EVT | 90 days post-EVT
  The rate of functional independence at 90 days post-EVT
The mortality rate within 90 days post-EVT | 90 days post-EVT
  The mortality rate within 90 days post-EVT

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai